CLINICAL TRIAL: NCT03299491
Title: An Implementation Study of Interventions to Promote Safe Motherhood in Jimma Zone Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Jimma University (Other); Ethiopian Ministry of Health, Jimma Zone (Unknown)
Responsible Party: Principal Investigator, Manisha Kulkarni, PhD, Assistant Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 108028-002
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Maternal Mortality; Maternal Morbidity
Keywords: Maternity Waiting Area; Ethiopia; Community Leader; Religious Leader; Skilled birth attendance; Postnatal care; Information, Education, Communication; Safe Motherhood; Health Extension Worker; Antenatal Care
MeSH Terms: conditions — Maternal Death; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MWA+IEC intervention (Experimental)
  Interventions: Other: MWA intervention; Other: IEC intervention
- IEC intervention (Experimental)
  Interventions: Other: IEC intervention
- Control (No Intervention)

INTERVENTIONS:
Other: MWA intervention — The MWA intervention will involve upgrading existing maternity waiting areas to ensure that essential supplies and services are available to create a comfortable environment for women to temporarily reside in and have easy access to skilled obstetric services.
  Arms: MWA+IEC intervention
Other: IEC intervention — Community and religious leaders will each attend one-day workshops designed using participatory, adult learning methods to help participants better understand the importance of maternal health care services, identify barriers to accessing care and to strategize how to promote utilization of services. Half-day workshops will conducted in subsequent years to build on shared experiences.
  Health extension workers will attend 3-day workshops to identify enablers and barriers to implementation of the safe motherhood components of the health extension program and strategize on how to engage community and religious leaders to support access to maternal health care services in their communities.
  Half-day workshops will conducted in subsequent years for each of the participant groups to build on shared experiences.
  Arms: IEC intervention; MWA+IEC intervention

SUMMARY:
Ethiopia has one of the highest rates of maternal mortality among all countries in Africa and indeed worldwide, with a maternal mortality ratio of 676 per 100,000 live births in 2011 (UNFPA, 2012). The majority of maternal deaths are preventable through early detection and management of complications, and access to adequate obstetric care (Say et al, 2014). However, in 2011 only 34% of women received antenatal care, 10% of births were delivered at a health facility and 7% of women received postnatal care during the first two days after delivery (Ethiopian DHS, 2011). Large distances and poor access to transport are two major obstacles that women face when trying to access services. In order to facilitate timely access to obstetric care, the Ethiopian Government introduced Maternity Waiting Areas (MWAs) at health centres to enable women to stay close to health facilities as they await delivery. Utilization of MWAs has generally been low due to the poor state of the homes and lack of adequate community support. This study aims to evaluate the effectiveness of two interventions to promote safe motherhood in increasing coverage of maternal health care services: (i) upgraded MWAs (ii) community and religious leader sensitization using information, education and communication (IEC) materials. The IEC materials are expected to increase leader awareness and support of antenatal care, facility deliveries, postnatal care and MWA use. Together with increased use of functional MWAs, improved support from leaders is expected to increase the proportion of facility-based births in interventions area. The interventions are also expected to positively impact antenatal care and postnatal care use in the study districts.

DETAILED DESCRIPTION:
A three-arm cluster trial design will be used to measure the impact of the intervention packages in three districts (Gomma, Seka Chekorsa, Kersa) in Jimma Zone, Ethiopia. Twenty-four clusters with 160 individuals each are required to detect a 17% change in the primary outcome (proportion of facility-based births) with 80% power,assuming a cluster autocorrelation of 0.8 and an intra-cluster correlation coefficient of 0.1. Primary health care units (PHCU) which consist of a health centre and several community-based health posts will serve as trial clusters. All PHCUs with maternity waiting areas (MWAs) constructed will be eligible for selection. Eligible women will be randomly selected from PHCU catchment areas stratified by MWA functionality and health centre basic emergency obstetric care (BEmOC) capacity. This is to ensure balanced distribution of poorly functioning MWAs and facilities with diminished BEmOC capacity between trial arms.

Cross-sectional household surveys will be conducted with eligible women to collect information on socio-demographics, knowledge, attitudes and practices regarding maternal health services, reproductive history and maternal health service utilization. Surveys will be administered by trained interviewers on tablet computers programmed using Open Data Kit at baseline prior to intervention roll out and at endline. Multilevel regression models will be used to quantify the effect of the intervention packages on outcomes of interest. Random effect terms for PHCUs will be included to account for the clustered nature of the data.

ELIGIBILITY:
Inclusion Criteria:

* Women who were pregnant up to one year prior to the baseline survey and had a live birth, stillbirth or abortion (spontaneous or induced) and are residents in the study districts during the survey period are eligible to take part in the study.

Exclusion Criteria:

* Women who are not able to provide informed consent due to severe illness or mental health conditions.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3784 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Facility-based birth coverage | Information on the primary outcome will be collected through surveys at baseline (prior to intervention roll out) and endline (approximately one and a half years after intervention roll out has commenced)
  Proportion of women who report giving birth to their last child at a health facility (health centre or hospital) which has skilled birth attendants present (doctor, midwife, clinical nurse).

SECONDARY OUTCOMES:
Antenatal care coverage | Information on secondary outcomes will be collected through surveys at baseline (prior to intervention roll out) and endline (approximately one and a half years after intervention roll out has commenced)
  Proportion of women who report making at least one antenatal care visit to a health facility during their last pregnancy.
Postnatal care coverage | Information on secondary outcomes will be collected through surveys at baseline (prior to intervention roll out) and endline (approximately one and a half years after intervention roll out has commenced)
  Proportion of women who report receiving a checkup from a healthcare worker at least once during the 42 days after delivery of their last child.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Kulkarni, PhD, Principal Investigator — University of Ottawa; Lakew Abebe, MPH, Principal Investigator — Jimma University

REFERENCES:
- [Result] Kurji J, Gebretsadik LA, Wordofa MA, Morankar S, Bedru KH, Bulcha G, Bergen N, Kiros G, Asefa Y, Asfaw S, Mamo A, Endale E, Thavorn K, Labonte R, Taljaard M, Kulkarni MA. Effectiveness of upgraded maternity waiting homes and local leader training on improving institutional births: a cluster-randomized controlled trial in Jimma, Ethiopia. BMC Public Health. 2020 Oct 22;20(1):1593. doi: 10.1186/s12889-020-09692-4. PMID 33092565
- [Derived] Kurji J, Kulkarni MA, Gebretsadik LA, Wordofa MA, Morankar S, Bedru KH, Bulcha G, Thavorn K, Labonte R, Taljaard M. Effectiveness of upgraded maternity waiting homes and local leader training in improving institutional births among women in the Jimma zone, Ethiopia: study protocol for a cluster-randomized controlled trial. Trials. 2019 Dec 4;20(1):671. doi: 10.1186/s13063-019-3755-z. PMID 31801584